CLINICAL TRIAL: NCT03901898
Title: Feasibility of an Implementation Intervention to Increase Attendance at Diabetic Retinopathy Screening: Protocol for a Cluster Randomised Pilot Trial
Brief Title: Feasibility of an Intervention to Increase Diabetic Retinopathy Screening Attendance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Dr Sheena McHugh, Principal Investigator, University College Cork
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: UCCork_IDEAs
Record Dates: First submitted 2019-03-28; First posted 2019-04-03 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Diabetes; Retinopathy
Keywords: screening; primary care; general practice; feasibility
MeSH Terms: conditions — Diabetes Mellitus; Retinal Diseases | interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: Four practices will be randomly assigned to the intervention group, while the other four practices will be assigned to the wait list control group. The wait list control group will deliver care as usual, and deliver the intervention after six months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training, audit, and reminders (Experimental): An investigator will deliver a 20-30-minute briefing on intervention delivery to all staff at participating practices, followed by one-on-one audit training (1 hour) with the staff member responsible for conducting the audit. Each practice conducts an audit of their patients with diabetes to identify all people who have not attended retinopathy screening with the national programme. At 6 months, practices conducts a re-audit. Practice staff add electronic alerts to the records of eligible patients, to prompt GPs and nurses to remind patients. Practices are reimbursed at study entry with further payment following intervention cessation based on number of patients audited. Face-to-face verbal reminders are delivered by GPs and practice nurses to eligible patients attending for an appointment during the study period. All eligible patients receive a reminder phone call from a practice nurse and a GP-endorsed reminder letter accompanied by an information leaflet.
  Interventions: Behavioral: Training, audit, and reminders
- Wait list control (Other): In control practices, the intervention will be delivered after 6 months. For the audit, administrators or practice nurses will use date restricted data extraction from the electronic medical record to capture data for the 12-month period prior to the intervention (study baseline) and 6 months after the study intervention period, during which they will have acted as control practices (follow-up). This will satisfy the baseline data collection prior to the delivery of the intervention to this group on study completion. This approach was chosen as collecting data at baseline (i.e. 6 months before intervention start) would constitute an intervention in those practices; knowledge of non-attenders would lead to a change in usual care as the control group would likely follow up patients immediately. Control practices will receive the same supports and training as intervention practices.
  Interventions: Behavioral: Intervention after 6 months (wait list)

INTERVENTIONS:
Behavioral: Training, audit, and reminders — Briefing and training for participating practices, baseline practice audit, addition of electronic prompts to patient records, GP-endorsed patient reminders (in person, phone and letter), and re-audit at 6 months.
  Arms: Training, audit, and reminders
Behavioral: Intervention after 6 months (wait list) — After 6 months, practices receive the intervention: briefing and training for participating practices, baseline practice audit, addition of electronic prompts to patient records, GP-endorsed patient reminders (in person, phone and letter).
  Arms: Wait list control

SUMMARY:
The purpose of this study is to test a way to support practices to improve attendance at retinopathy screening among people with diabetes. This new approach will be delivered to staff in general practice and involves: 1) briefing and audit training for practice staff; 2) electronic alerts on patient files to prompt GPs and nurses to remind patients, 3) face-to-face, phone and letter reminders and a brief information sheet for people with diabetes who have not attended screening, and; 4) payment to practices. The practice will carry out an audit to identify patients who have not attended screening, and re-audit at 6 months to identify any changes in attendance. The study will test this new approach over six months in eight different practices to determine whether it is feasible to deliver in a real-world setting. Four practices will be randomly assigned to receive the new approach straight away (intervention group), while the other four practices will be assigned to the group who wait, deliver care as usual, and roll out the new approach after six months (wait-list-control group). After the new approach has been tested for six months, the research team will use staff questionnaires, and carry out focus groups and interviews with patients and practice staff to learn about their experiences. The time and resources needed to deliver the approach will also be recorded to estimate the cost of delivering the new approach and how feasible it would be to carry out a larger study.

DETAILED DESCRIPTION:
Aims and objectives.

The current study will address uncertainties about feasibility, economic evaluation, and the study procedures. The feasibility pilot study is needed to determine whether a larger-scale trial would be viable. Specifically, it will address the questions:

1. Are the intervention content, delivery and procedures acceptable to people with diabetes who will receive the intervention, and staff who will deliver the intervention?
2. Are the data collection processes, including mode and duration of data collection and outcome measures used, acceptable to staff?
3. Is the intervention feasible to deliver in primary care practice, in terms fidelity of delivery and receipt of the intervention?
4. Is the study feasible in terms of recruitment and retention procedures and data collection?
5. What are the costs associated with the intervention?

Intervention. The intervention involves components which target practice staff (1. brief training 2. electronic prompt, and 3. reimbursement) and components which target patients with type 1 or type 2 diabetes who have not attended screening (1. face-to-face reminder message and information leaflet; 2. phone reminder; 3. GP-endorsed reminder letter and information leaflet). The intervention will be delivered over 6 months. The practice will conduct an audit of their patients with diabetes at baseline and re-audit at 6 months. Only practice staff will access patient files for the purpose of the audit. Only practice staff will have contact with patients during intervention delivery; a member of the practice team will issue the face-to-face, phone and letter reminders.

Methods. IDEAs (Improving Diabetes Eye-screening Attendance) is a cluster randomised feasibility pilot trial, including an embedded process evaluation and economic evaluation. In the current study, general practices will be randomly allocated to intervention or wait-list control groups following stratification by practice size (i.e. single/two-handed or group practice (3 more or GPs). Practices in the wait-list control group will receive the same intervention at 6 months. A multi-method approach will be used to evaluate the trial and study procedures, and to examine the acceptability and feasibility of the intervention from the perspective of practice staff and patients. Quantitative and qualitative data will be collected on intervention delivery, research processes, and implementation outcomes. Data will be collected at the practice, health professional and patient level. Data will be collected by practice staff and study researchers during intervention delivery. An economic evaluation will be conducted to estimate the cost of delivering the intervention in general practice

ELIGIBILITY:
Inclusion Criteria (practices):

* Computerised record system
* Practice nurse

Inclusion Criteria (patients)

* 18 years or over
* Diagnosed diabetes (type 1 or type 2)
* Has been audited as part of the practice-level intervention
* Eligible to attend the national screening programme but has not registered, consented to, and attended the programme.

Exclusion Criteria (patients):

• Has retinopathy and are currently under surveillance or receiving treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2020-10-12 (Actual); Study Completion 2020-10-12 (Actual)

PRIMARY OUTCOMES:
Number of patients who intend to contact RetinaScreen | 6 months
  Patient self-report during phone call from the practice
Number of patients who have contacted the national screening programme | 6 months
  Patient self-report during phone call from the practice
Number of patients who have attended screening | 6 months
  Number obtained from practice electronic health records. Letter received from the national screening programme on patient record.

CONTACTS AND LOCATIONS:
Overall Officials: Sheena M McHugh, PhD, Principal Investigator — University College Cork
Locations (1):
- University College Cork, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tracey ML, McHugh SM, Fitzgerald AP, Buckley CM, Canavan RJ, Kearney PM. Trends in blindness due to diabetic retinopathy among adults aged 18-69years over a decade in Ireland. Diabetes Res Clin Pract. 2016 Nov;121:1-8. doi: 10.1016/j.diabres.2016.08.016. Epub 2016 Aug 30. PMID 27612011
- [Background] Lawrenson JG, Graham-Rowe E, Lorencatto F, Burr J, Bunce C, Francis JJ, Aluko P, Rice S, Vale L, Peto T, Presseau J, Ivers N, Grimshaw JM. Interventions to increase attendance for diabetic retinopathy screening. Cochrane Database Syst Rev. 2018 Jan 15;1(1):CD012054. doi: 10.1002/14651858.CD012054.pub2. PMID 29333660
- [Background] Zhang X, Norris SL, Saadine J, Chowdhury FM, Horsley T, Kanjilal S, Mangione CM, Buhrmann R. Effectiveness of interventions to promote screening for diabetic retinopathy. Am J Prev Med. 2007 Oct;33(4):318-35. doi: 10.1016/j.amepre.2007.05.002. PMID 17888859
- [Derived] Riordan F, Murphy A, Dillon C, Browne J, Kearney PM, Smith SM, McHugh SM. Feasibility of a multifaceted implementation intervention to improve attendance at diabetic retinopathy screening in primary care in Ireland: a cluster randomised pilot trial. BMJ Open. 2021 Oct 19;11(10):e051951. doi: 10.1136/bmjopen-2021-051951. PMID 34667010
- [Derived] Riordan F, Racine E, Smith SM, Murphy A, Browne J, Kearney PM, Bradley C, James M, Murphy M, McHugh SM. Feasibility of an implementation intervention to increase attendance at diabetic retinopathy screening: protocol for a cluster randomised pilot trial. Pilot Feasibility Stud. 2020 May 12;6:64. doi: 10.1186/s40814-020-00608-y. eCollection 2020. PMID 32426158